CLINICAL TRIAL: NCT01278511
Title: A Prospective Pilot Study Validating the Canadian C-Spine Rule in a Pre-hospital Setting
Brief Title: Prospective Pilot Study Validating the Canadian C-Spine Rule Pre-hospital
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Pieter Jan Van Asbroeck, Dr. Pieter Jan Van Asbroeck, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S52940
Record Dates: First submitted 2011-01-13; First posted 2011-01-19 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Injury of Cervical Spine; Cervical Spine Fractures
Keywords: Canadian C-Spine Rule; Prehospital Emergency Care; Cervical Spine Injuries; Cervical Spine Fractures; Emergency Medicine Undergraduates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canadian C-Spine Rule (Experimental)
  Interventions: Other: Canadian C-Spine rule

INTERVENTIONS:
Other: Canadian C-Spine rule — Emergency medicine undergraduates will accompany prehospital emergency crews and apply the Canadian C-Spine rule, though cervical collar will be applicated per current protocol.

SUMMARY:
This study is designed to evaluate the safety, level of performance and level of comfort with the Canadian C-Spine rule in a prehospital setting by emergency medicine undergraduates.

ELIGIBILITY:
Inclusion Criteria:

* Alert, stable, adult patients presenting with an acute possible injury to the cervical spine
* Alert: GCS ≥ 14
* Stable:

  * systolic blood pressure ≥ 90 mmHg
  * respiratory frequency 12 - 20 / min
  * adult ≥ 18 years old
* Acute: ≤ 4
* Possible injury to the cervical spine:

  * posterior neck pain following any mechanism
  * no neck pain but visible injury above the clavicles
  * no neck pain or visible injury above the clavicles but a mechanism that indicates a cervical spine injury

Exclusion Criteria:

* Acute paralysis (quadriplegia, paraplegia)
* Penetrating trauma to the neck
* Patients with known vertebral disease (ankylosing spondylitis, rheumatoid arthritis, spinal stenosis, or previous cervical spine surgery)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Missed cervical spine injuries and fractures | At the first visit to the emergency department until 30 days after inclusion

SECONDARY OUTCOMES:
Performance of the Canadian c-spine rule | Analyzed at the end of the pilot study in april 2011
  Performance includes rule accuracy
Level of comfort | Analyzed at the end of the pilot study in april 2011
  Level of comfort with the decision of the canadian c-spine rule as this is important for a possible implication in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Koen Bronselaer, MD, PhD, Study Director — Emergency Department of the University Hospitals, Catholic University Leuven; Marc Sabbe, MD, PhD, Principal Investigator — Emergency Department of the University Hospitals, Catholic University Leuven; Pieter Jan Van Asbroeck, Drs, Principal Investigator — Emergency Department of the University Hospitals, Catholic University Leuven
Locations (1):
- Emergency Department of the University Hospitals, Catholic University Leuven, Leuven, Vlaams-Brabant, Belgium